CLINICAL TRIAL: NCT06867003
Title: Effectiveness of Physical Therapy With &Amp; Without Bracing on Posture, Pain and Functional Outcomes in Office Workers With Kyphosis
Brief Title: Comparison of Exercise With & Without Bracing in Office Workers With Kyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-01009 Yasir Khan
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Kyphosis
Keywords: Kyphosis
MeSH Terms: conditions — Kyphosis | interventions — Physical Therapy Modalities; Braces; Exercise

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Masking Description: this study follows an analytical research model designed to compare effectiveness of Physical Therapy with and without Bracing on Posture, Pain, and Functional Outcomes in Office Workers with Kyphosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy with bracing (Experimental): Effectiveness of physical therapy with bracing
  Interventions: Other: physical therapy with bracing
- physical therapy without bracing (Placebo Comparator): Effectiveness of physical therapy without bracing
  Interventions: Other: physical therapy without bracing

INTERVENTIONS:
Other: physical therapy with bracing — Strengthens the upper back muscles and reduces tension:
  1. Stand or sit with an upright posture and shoulders pulled back
  2. Squeeze your shoulder blades together as tightly as you can and hold for five to ten seconds
  Other Names: Exercise
  Arms: Physical therapy with bracing
Other: physical therapy without bracing — Strengthens the upper back muscles and reduces tension:
  1. Stand or sit with an upright posture and shoulders pulled back
  2. Squeeze your shoulder blades together as tightly as you can and hold for five to ten seconds
  Arms: physical therapy without bracing

SUMMARY:
The study aims to Compare PT and bracing in improving posture, pain, and functionality in patient with kyphosis.

It also assess the additive benefits of combining PT with bracing. It also identify sustainable, non-surgical approaches for managing kyphosis in office

DETAILED DESCRIPTION:
The study focuses on understanding Kyphosis, defined as excessive forward curvature of the thoracic spine, has become increasingly prevalent in modern work environments due to the sedentary nature of desk jobs. Kyphosis, characterized by a rounded upper back or "hunchback" appearance, is a clinical and postural problem with significant physical, functional, and psychosocial implications. Among office workers, the condition is primarily postural, driven by long hours of desk work, inappropriate ergonomic settings, and inadequate postural awareness. The increasing prevalence of kyphosis in this demographic has led to a pressing need for effective nonsurgical management strategies, including physical therapy (PT) and spinal bracing.

ELIGIBILITY:
Inclusion Criteria:

* Office workers diagnosed with Postural Kyphosis
* age limit 30 to 45years
* Experience of upper back or neck pain lasting at least three months
* Spend a minimum of 6 hours per day in a seated position for work.

Exclusion Criteria:

* History of spinal surgery, severe scoliosis, or other significant spinal deformities.

Current engagement in any structured physical therapy program or use of bracing for posture. Any neurological or musculoskeletal disorders impacting posture or movement.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 4 weeks
  The questionnaire consists of 10 sections, each with 6 response options (scored 0 to 5). If all 10 sections are completed, the maximum score is 50.
Visual Analogue Scale (VAS) | 4 weeks
  A 10 cm horizontal line with "No Pain" (0) on the left and "Worst Pain" (10) on the right.

CONTACTS AND LOCATIONS:
Overall Officials: Ataur Rahman, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University malakand campus, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No